CLINICAL TRIAL: NCT01072266
Title: A Phase 1, Open-label, Dose-Escalation Study to Determine the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of INCB028060 in Subjects With Advanced Malignancies
Brief Title: A Dose-escalation Study in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 28060-101
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Solid Tumor; Advanced Cancer; Metastatic Cancer
Keywords: Refractory, Advanced malignancies
MeSH Terms: conditions — Neoplasm Metastasis | interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INCB028060 (Experimental): Subjects will be enrolled and treated in cohorts of three and each observed a minimum of 28 days before the next group of patients may be enrolled and receive study drug. The initial cohort will be treated with 10 mg QD. The second cohort will be treated with 20 mg QD. The third cohort will be treated with 50 mg QD. Subsequent cohorts will be treated with two times the dose of the prior cohort to a limited toxicity level.
  Interventions: Drug: INCB028060

INTERVENTIONS:
Drug: INCB028060 — 10 mg and 50 mg capsules will be provided and dosed per the dosing schedule.

SUMMARY:
This is an open label, dose escalation study using a 3 + 3 design to determine if INCB028060 (study drug) is safe, well-tolerated and effective in patients with advanced malignancies. Patients will be enrolled and treated in cohorts of three and each observed a minimum of 28 days before the next group is enrolled and may begin to receive study drug. Doses will be escalated unless a dose-limiting toxicity (DLT) is observed in one of three subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with neoplastic disease refractory to currently available therapies or for which no effective treatment is available
* Subjects with life expectancy of 12 weeks or longer.
* Subjects with Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

Exclusion Criteria:

* Subjects who received any anti-cancer medications in the 21 days prior to receiving their first dose of study medication or 6 weeks for mitomycin-C or nitrosoureas.
* Subjects with history of brain metastases or spinal cord compression.
* Subjects who have undergone a bone marrow or solid organ transplant.
* Subjects who have had major surgery within 4 weeks prior to study entry or had minor surgical procedure within 7 days prior to initiating treatment.
* Subjects with clinically significant non-healing or healing wounds or subjects with lung tumor lesions with increased likelihood of bleeding
* Subjects with a history of any gastrointestinal condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be the primary endpoint and will be assessed by monitoring the frequency, duration, and severity of AEs | Baseline and every 1-2 weeks based on protocol visit schedule until the end of study or early termination visit.

SECONDARY OUTCOMES:
c-MET inhibitory activity determined by the relationship between blood levels of INCB028060 and the percent inhibition of c-MET phosphorylation | Predose, specific hours post-dose on day and Day 15 of Cycle 1.
  Samples will be collected at 0 (predose) and 2, 4, and 6 hours after dosing on Day 1 and Day 15 of Cycle 1 for subjects undergoing full PK analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, Study Director — Incyte Corporation
Locations (2):
- United States (2):
  - Baltimore, Maryland
  - Nashville, Tennessee